CLINICAL TRIAL: NCT05322759
Title: Comparison of Halliwick Exercises and Aquatic Excercices on Gross Motor Function, Trunk Stability and Hand Function in Spastic CP
Brief Title: Halliwick and Aquatic Exercises in Spastic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU Nimra Arif
Record Dates: First submitted 2022-01-24; First posted 2022-04-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Spastic Cerebral Palsy
Keywords: Halliwick exercises; Aquatic exercises; Gross Motor Function measurment; Trunk control
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aquatic exercises (Active Comparator): this group receives sessions for consecutive 8 weeks and 3 days per week. warm up for 10 min, that will include walking in shallow water and stretchings of upper and lower extremities. After that APE for 30 min followed cool down period for 5 min. exercise frequency is 3 sets of each exercise with 15 repetitions.
  Interventions: Other: aquatic exercises; Other: halliwick exercise programme
- Halliwick exercise programme (Experimental): this group receives sessions for consecutive 8 weeks and 3 days per week. warm up for 10 min that specifically includes mental adjustments along with walking in shallow side of pool and static stretchings. After that Halliwick exercise programme for 30 min that followed by cool down period for 5 min. exercise frequency is 3 sets of each exercise with 15 repetitions.
  Interventions: Other: aquatic exercises; Other: halliwick exercise programme

INTERVENTIONS:
Other: aquatic exercises — aquatic polymetric exercises for 30 min including hip abduction/adduction, knee flexion/extension, hip flexion/extension, holding pool from sides, bending forward and picking up objects, shoulder flexion/extension kangroo jumpes, jumping to sides.
Other: halliwick exercise programme — Halliwick exercise programme for 30 min include sagittal rotations, transversal rotations, longitudnal rotations and combined rotations.

SUMMARY:
The aim of this research is to find and compare the effects of halliwick exercises and aquatic exercises on gross motor function, trunk stability and hand function in spastic cerebral palsy.

DETAILED DESCRIPTION:
Randomized controlled trials done at Dream Child institute and Children hospital complex Multan. The sample size was 32. The subjects were divided in two groups, 16 subjects in halliwick exercise group and 20 in aquatic exercise group. Study duration was of 6 months. Sampling technique applied was convenient non probability sampling technique. Only 13-16 years diagnosed spastic cerebral pals individuals were included. Tools used in the study are Gross motor function measure (GMFM-66), Trunk impairment scale (TIS) and Nine-hole peg test (NHPT). Data was being analyzed through SPSS 22.

ELIGIBILITY:
Inclusion Criteria:

* Both genders Male & female
* Age 13-16 years
* Able to use assistive devices
* Diagnosed CP children
* Able to follow verbal commands

Exclusion Criteria:

* Unstable seizures

  * had a surgery for the last 12 months or receive medication for spasticity
  * Associated cognitive issue
  * Incontinence
  * Persistent infection

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
GMFM-88 | first reading at 0 week
  It is an observational clinical measure designed to evaluate gross motor function in children with cerebral palsy.
GMFM-88 | final reading at 8 week
  It is an observational clinical measure designed to evaluate gross motor function in children with cerebral palsy.
Trunk Impairment Scale | First reading at 0 week
  this scale measures static sitting and dynamic balance as well as trunk co-ordination. this aims to score the quality of trunk movement and to be as a guide for treatment.
Trunk Impairment Scale | Final reading at 8 week
  this scale measures static sitting and dynamic balance as well as trunk co-ordination. this aims to score the quality of trunk movement and to be as a guide for treatment.
Nine Hole Peg Test | first reading at 0 week
  it is a standerized test for measuring hand function and finger dexterity. scoring is done on the basis of average time for consecutive 4 trial with dominant hand and then by non-dominant hand.
Nine Hole Peg Test | final reading at 8 week
  it is a standerized test for measuring hand function and finger dexterity. scoring is done on the basis of average time for consecutive 4 trial with dominant hand and then by non-dominant hand.

CONTACTS AND LOCATIONS:
Overall Officials: Binash Afzal, Phd*, Principal Investigator — Riphah International University
Locations (1):
- Binash Afzal, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gurpinar B, Kara B, Idiman E. Effects of aquatic exercises on postural control and hand function in Multiple Sclerosis: Halliwick versus Aquatic Plyometric Exercises: a randomised trial. J Musculoskelet Neuronal Interact. 2020 Jun 1;20(2):249-255. PMID 32481240
- [Background] Akinola BI, Gbiri CA, Odebiyi DO. Effect of a 10-Week Aquatic Exercise Training Program on Gross Motor Function in Children With Spastic Cerebral Palsy. Glob Pediatr Health. 2019 Jun 25;6:2333794X19857378. doi: 10.1177/2333794X19857378. eCollection 2019. PMID 31263742
- [Background] Adar S, Dundar U, Demirdal US, Ulasli AM, Toktas H, Solak O. The effect of aquatic exercise on spasticity, quality of life, and motor function in cerebral palsy. Turk J Phys Med Rehabil. 2017 Aug 14;63(3):239-248. doi: 10.5606/tftrd.2017.280. eCollection 2017 Jun. PMID 31453460
- [Background] Ballington SJ, Naidoo R. The carry-over effect of an aquatic-based intervention in children with cerebral palsy. Afr J Disabil. 2018 Oct 29;7(0):361. doi: 10.4102/ajod.v7i0.361. eCollection 2018. PMID 30473998
- [Background] Terrens AF, Soh SE, Morgan P. The safety and feasibility of a Halliwick style of aquatic physiotherapy for falls and balance dysfunction in people with Parkinson's Disease: A single blind pilot trial. PLoS One. 2020 Jul 30;15(7):e0236391. doi: 10.1371/journal.pone.0236391. eCollection 2020. PMID 32730325
- [Background] Veldema J, Jansen P. Aquatic therapy in stroke rehabilitation: systematic review and meta-analysis. Acta Neurol Scand. 2021 Mar;143(3):221-241. doi: 10.1111/ane.13371. Epub 2020 Nov 22. PMID 33141446
- [Background] Carayannopoulos AG, Han A, Burdenko IN. The benefits of combining water and land-based therapy. J Exerc Rehabil. 2020 Feb 26;16(1):20-26. doi: 10.12965/jer.1938742.371. eCollection 2020 Feb. PMID 32161731
- [Background] Perez-de la Cruz S. Effect of an Aquatic Balance-Training Program in Patients with Chronic Stroke: A Single-Group Experimental Pilot Study. Medicina (Kaunas). 2020 Nov 28;56(12):656. doi: 10.3390/medicina56120656. PMID 33260785